CLINICAL TRIAL: NCT04817683
Title: Exploration of the Relationship Between Mobile Phone Addiction and Functional Gastrointestinal Disorders, a Cross-sectional Study
Brief Title: Study on the Relationship Between Mobile Phone Addiction and Functional Gastrointestinal Disorders
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020024
Record Dates: First submitted 2020-07-03; First posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: IBS - Irritable Bowel Syndrome
Keywords: IBS，FD，MPA
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross-sectional study was conducted to collect the relevant data of college students' mobile phone addiction and FGIDs (IBS, FD) in the form of questionnaire, so as to understand the situation of college students' mobile phone addiction and the incidence of FGIDs (IBS and FD), and explore the correlation, so as to provide new ideas and scientific basis for the prevention, diagnosis and treatment of FGIDs among college students.

DETAILED DESCRIPTION:
This study adopts the method of cross-sectional survey to collect the relevant data of Chinese college students' mobile phone addiction and FGIDs (IBS, FD) in the form of online and face-to-face questionnaire, so as to understand the situation of Chinese college students' mobile phone addiction and the incidence of FGIDs (IBS, FD), and explore the correlation, so as to provide new ideas and scientific basis for the prevention, diagnosis and treatment of FGIDs.

ELIGIBILITY:
Inclusion Criteria:

* College students from all over the country, over 17 years old, have a physical examination before entering school
* Sign the informed consent form, voluntarily participate and fill in the questionnaire

Exclusion Criteria:

* People with diabetes, hyperthyroidism or hypothyroidism, peptic ulcer, inflammatory bowel disease, digestive tract tumor or severe medical and surgical disease
* History of abdominal surgery (such as esophagus, stomach, small intestine, colon, rectum, appendix, gallbladder, hysterectomy, cesarean section)
* Recently, there are some alarm symptoms, such as relieving black stool, bloody stool, hematemesis, abnormal anemia, fever, abnormal weight loss (no intention to lose weight, weight loss 5 kg in 3 months), change of defecation habits, dysphagia and so on
* In the past 4 weeks, he has taken drugs that affect the judgment of gastrointestinal symptoms, such as anti-inflammatory painkillers, diazepam drugs, anti-anxiety drugs, depressants and so on

Min Age: 17 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: College students over the age of 17 across the country
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2020-12-28 (Actual)

PRIMARY OUTCOMES:
Incidence of irritable bowel syndrome among College Students.Risk factors of irritable bowel syndrome. | 2020.07.03-2020.12.28
  The irritable bowel syndrome was diagnosed by the Rome IV diagnostic questionnaire, and then the incidence of irritable bowel syndrome was calculated by SPSS. Through PHQ-9 questionnaire to diagnose depression, GAD-7 questionnaire to diagnose anxiety, MPAI questionnaire to diagnose mobile phone addiction, AIS questionnaire to diagnose insomnia, logistic regression analysis to calculate OR value and P value, to understand the relationship between irritable bowel syndrome and anxiety, depression, insomnia, mobile phone addiction.

SECONDARY OUTCOMES:
Incidence of functional dyspepsia among College Students.Risk factors of functional dyspepsia. | 2020.07.03-2020.12.28
  The functional dyspepsia was diagnosed by the Rome IV diagnostic questionnaire, and then the incidence of functional dyspepsia was calculated by SPSS. Through PHQ-9 questionnaire to diagnose depression, GAD-7 questionnaire to diagnose anxiety, MPAI questionnaire to diagnose mobile phone addiction, AIS questionnaire to diagnose insomnia, logistic regression analysis to calculate OR value and P value, to understand the relationship between functional dyspepsia and anxiety, depression, insomnia, mobile phone addiction.

CONTACTS AND LOCATIONS:
Overall Officials: Jinhai Wang, MD, Study Director — Second Affilated Hospital of Xi'an Jiaotong University
Locations (1):
- The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No